CLINICAL TRIAL: NCT04398953
Title: A Single-arm, Multicenter Phase II Clinical Trial of TQ-B3525 Tablet in the Treatment of Relapsed / Refractory Mantle Cell Lymphoma (MCL)
Brief Title: A Study of TQ-B3525 Tablet in the Treatment of Relapsed / Refractory Mantle Cell Lymphoma (MCL)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQ-B3525-II-02
Record Dates: First submitted 2020-05-19; First posted 2020-05-22 (Actual); Last update posted 2020-09-11 (Actual); Status verified 2020-01

CONDITIONS: Relapsed / Refractory Mantle Cell Lymphoma (MCL)
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — TQ-B3525

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TQ-B3525 tablet (Experimental): TQ-B3525 tablet administered orally.
  Interventions: Drug: TQ-B3525

INTERVENTIONS:
Drug: TQ-B3525 — TQ-B3525 tablet administered 20mg orally, once daily in 28-day cycle.

SUMMARY:
This is a study to evaluate the safety and efficacy of TQ-B3525 tablets in patients with relapsed / refractory mantle cell lymphoma (MCL).

ELIGIBILITY:
Inclusion Criteria:

* 1. Understood and signed an informed consent form; 2. Eastern Cooperative Oncology Group (ECOG) performance status score of 0 to 2; Life expectancy ≥ 3 months; 3. Relapsed / refractory MCL; 4. Has received at least one-line and less than four lines of previous treatment, the latest treatment confirmed no objective response, or disease progress after treatment; 5. Has at least one measurable lesion; 6. Adequate organ system function; 7. Male or female subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 6 months after the last dose of study (such as intrauterine devices , contraceptives or condoms) ；No pregnant or breastfeeding women, and a negative pregnancy test are received within 7 days before the first administration.

Exclusion Criteria:

* 1. Has central nervous system violation; 2. Has received other PI3K inhibitors; 3. Has diagnosed and/or treated additional malignancy within 3 years prior to the first administration; 4. Has history of interstitial lung disease; 5. Has a history of immunodeficiency diseases; 6. Has multiple factors affecting oral medication; 7. Has adverse events caused by previous therapy except alopecia that did not recover to ≤grade 1; 8. Has received systemic steroid treatment within 7 days before the first administration; 9. Has received other systemic anti-tumor medications within 4 weeks before the first administration, or still within the 5 half-life of the medication, which occurs first; 10. Has palliative radiation therapy within 4 weeks before the first administration; 11. Has active infections within 4 weeks before the first administration; 12. Has received surgery, or unhealed wounds within 4 weeks before the first administration; 13. Has a history of autologous hematopoietic stem cell transplant within 6 months or allogeneic hematopoietic stem cell transplant; 14. QTCF > 480ms, LVEF < 50%; 15. Urinary protein ≥ 2 +, and urinary protein quantity >1.0 g in 24 hours within 7 days; 16. Has active hepatitis B or C; 17. Has psychotropic substances abuse or a mental disorder; 18. Has other conditions that make it inappropriate for the patient to be enrolled based on investigator's opinion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2020-07-20 (Actual); Primary Completion 2021-09 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) assessed by Independent Review Committee (IRC) | up to 12 months
  Percentage of subjects achieving complete response (CR) and partial response (PR) based on investigator.

SECONDARY OUTCOMES:
Disease control rate（DCR） | up to 12 months
  Percentage of subjects achieving complete response (CR) and partial response (PR) and stable disease (SD).
Duration of Response (DOR) | up to 12 months
  DOR defined as time from earliest date of disease response to earliest date of disease progression based on radiographic assessment.
Progression-free survival (PFS) | up to 12 months
  PFS was defined as the time from the date of study enrollment to the date of the first of the following events, objective disease progression or death due to any cause.
Overall survival (OS) | up to 18 months
  OS defined as the time from the first dose to death from any cause. Survival time was censored at the date of last contact for patients who were still alive or lost to follow-up.
Biomarkers | up to 12 months
  To assess the changes of genes related to PI3K pathway and bypass in the tissues and / or plasma of enrolled patients.

CONTACTS AND LOCATIONS:
Locations (39):
- China (39):
  - Anhui Cancer Hospital, Hefei, Anhui
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Beijing Boren Hospital, Beijing, Beijing Municipality
  - Beijing Shijitan Hospital Affiliated to Capital Medical University, Beijing, Beijing Municipality
  - Cancer Hospital of Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - The Fifth Medical Center of PLA General Hospital, Beijing, Beijing Municipality
  - The Third Hospital of Peking University, Beijing, Beijing Municipality
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Union Hospital Affiliated to Fujian Medical University, Fuzhou, Fujian
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - The Second Hospital of Lanzhou University, Lanzhou, Gansu
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Guangxi Medical University Affiliated Tumor Hospital, Nanning, Guangxi
  - Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Hunan Cancer Hospital, Changsha, Hunan
  - Huai'an first people's Hospital, Huaian, Jiangsu
  - Jiangsu Cancer Hospital, Nanjing, Jiangsu
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - Nantong Tumor Hospital, Nantong, Jiangsu
  - The First Affiliated Hospital of Suzhou University, Suzhou, Jiangsu
  - Jiangxi Cancer Hospital, Nanchang, Jiangxi
  - The First Hospital of Jilin University, Changchun, Jilin
  - Affiliated Zhongshan Hospital of Dalian University, Dalian, Liaoning
  - The First Affiliated Hospital of Dalian Medical University, Dalian, Liaoning
  - The Second Affiliated Hospital of Dalian Medical University, Dalian, Liaoning
  - Affiliated Hospital of Binzhou Medical College, Binzhou, Shandong
  - Qingdao Central Hospital, Qingdao, Shandong
  - Weifang People's Hospital, Weifang, Shandong
  - Weihai Central Hospital, Weihai, Shandong
  - Weihai Municipal Hospital, Weihai, Shandong
  - Shanghai Tongji Hospital, Shanghai, Shanghai Municipality
  - Shanxi Provincial People's Hospital, Xi’an, Shanxi
  - Hematology Hospital of Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality
  - Tianjin Cancer Hospital, Tianjin, Tianjin Municipality
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - Tianjing People's Hospital, Tianjin, Tianjin Municipality